CLINICAL TRIAL: NCT04290520
Title: Optimization of Frozen Embryo Transfers by Studying Progesterone on the Day of Transfer
Acronym: OTEC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2020/SH-01
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Infertility; IVF
MeSH Terms: conditions — Infertility | interventions — Biological Assay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: bioassay — Serum progesterone level (ng/ml)

SUMMARY:
The number of embryo transfers after freezing has increased over the last 10 years due to improvements in embryo freezing techniques and in particular the development of vitrification. This has also been made possible by changes in clinical protocols favouring freezing in patients at high risk of hyperstimulation and by different methods of endometrial preparation to receive embryos after rewarming.

In fact, embryo transfer requires endometrial preparation to make implantation possible. There are various protocols for endometrial preparation. Endometrial preparations in the natural cycle, with or without induction of ovulation by FSH, require more regular monitoring, and allow the development of a main follicle that will give a corpus luteum that will secrete progesterone in the luteal phase, which can be supported by the supply of exogenous progesterone. In contrast, endometrial preparations in hormone replacement therapy (HRT) cycles are done by administering estradiol orally or transdermally to stimulate endometrial growth while blocking the patient's gonadotropic axis, and administering progesterone in the luteal phase to differentiate the endometrium. This preparation has the advantage of being simpler to monitor and organize.

There is currently no consensus on a type of preparation that would give better results, and although the literature seems to show that there would be more miscarriages in a substituted cycle, there does not seem to be any difference in the birth rate per cycle in the end, whatever the type of endometrial preparation.

Some teams have shown that in HRT, there appears to be more miscarriage when the progesterone level measured on the day of the frozen embryo transfer is lower, especially below a threshold of 9ng/mL. Labarta showed ESHRE in July 2019 that modifying the endometrial preparation if the progesterone level is below 9ng/mL on the day of transfer by adding subcutaneous progesterone (Progiron) resulted in a lower miscarriage rate, comparable to the usual miscarriage rates in spontaneous pregnancy.

Thus, if the miscarriage rate is higher in HRT than in the natural cycle, and if this is related to "luteal insufficiency" characterized by a lower circulating serum progesterone level, the hypothesis of this study in the investigator's population would be that the serum progesterone level on the day of the frozen embryo transfer would be lower in HRT than in the spontaneous cycle.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have benefited from a frozen embryo transfer during the inclusion period in the MPA centre of the CHU Caremeau Nimes are included.
* Adult patient (≥18 years of age) and under 43 years of age.

Exclusion Criteria:

* Patients who did not receive progesterone dosing on the day of transfer are excluded from the study.
* Patients who objected to the use of their data.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: These are MPA patients who have undergone embryo freezing and endometrial preparation for embryo replacement.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The main objective of our study is to compare progesterone levels on the day of embryo transfer according to the endometrial preparation protocol. | the day of the embryo transfer
  Serum progesterone level (ng/ml)

CONTACTS AND LOCATIONS:
Locations (1):
- CHUNimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No